CLINICAL TRIAL: NCT02233543
Title: A Multicenter, 4-week Crossover (Total Duration 12 Weeks), Placebo-controlled, Double-blind Study to Determine the Impact of QVA149 (Indacaterol/Glycopyrronium) 85/43 µg on Nocturnal Oxygen Levels in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Multicenter, 4-week Crossover (Total Duration 12 Weeks) to Determine the Impact of QVA149 on Nocturnal Oxygen Levels in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149ANO01
Record Dates: First submitted 2014-08-19; First posted 2014-09-08 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; QVA149; nocturnal oxygen levels; combination bronchodilator
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; indacaterol; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First QVA149 (indacaterol/glycopyrronium), then Placebo (Experimental): Participants received 4 weeks of QVA149 85/43 μg delivered dose once daily in the morning between 08:00 and 11:00 AM at approximately the same time every day followed by 2 weeks washout. Then participants received 4 weeks of placebo once daily in the morning between 08:00 and 11:00 AM at approximately the same time every day.
  Interventions: Drug: QVA149; Drug: QVA149 Placebo
- First Placebo, then QVA149 (indacaterol/glycopyrronium) (Experimental): Participants received 4 weeks of placebo once daily in the morning between 08:00 and 11:00 AM at approximately the same time every day followed by 2 weeks washout. Then participants received 4 weeks of QVA149 85/43 μg delivered dose once daily in the morning between 08:00 and 11:00 AM at approximately the same time every day.
  Interventions: Drug: QVA149; Drug: QVA149 Placebo

INTERVENTIONS:
Drug: QVA149 — Delivered once daily via single-dose dry powder inhaler
  Other Names: indacaterol/glycopyrronium,; Ultibro Breezhaler
Drug: QVA149 Placebo — Placebo delivered once daily via single-dose dry powder inhaler

SUMMARY:
The purpose of this study was to determine whether a fixed dose combination of indacaterol and glycopyrronium (QVA149) has an impact on night-time blood oxygen levels in Chronic Obstructive Pulmonary Disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD (according to GOLD guidelines, updated 2014) with a post-bronchodilator FEV1/FVC <0.70
* Patients with a post-bronchodilator FEV1 ≥30% and <60% of the predicted normal value
* Resting daytime oxygen saturation levels measured by pulse oximetry of ≤95% SpO2
* Smoking history of at least 10 pack years (Ten pack-years are defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years)

Exclusion Criteria:

* An exacerbation of COPD (treatment with oral or parenteral antibiotics and/or glucocorticosteroids and/or hospitalization related to COPD) within 4 weeks prior to screening or during the run-in period
* Diagnosed asthma
* Patients receiving regular long term oxygen therapy (LTOT)
* Ongoing / planned rehabilitation during the study period
* Three or more awakenings during the night leading to toilet visit or other reasons for exiting the bed during the last week prior to the screening visit due to non-COPD reasons

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-11-30 (Actual); Primary Completion 2016-06-26 (Actual); Study Completion 2016-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Hvidovre
- Novartis Investigative Site, Bergen, Norway
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio.
Period: Period 1
Arm/Group | First QVA149 (Indacaterol/Glycopyrronium), Then Placebo | First Placebo, Then QVA149 (Indacaterol/Glycopyrronium)
Started | 22 | 16
Completed | 19 | 13
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Participants required other treatment. | 2 | 3
Period: Period 2
Arm/Group | First QVA149 (Indacaterol/Glycopyrronium), Then Placebo | First Placebo, Then QVA149 (Indacaterol/Glycopyrronium)
Started | 19 | 13
Completed | 17 (1 participant erroneously received QVA149 during both periods.) | 12
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Participant required other treatment. | 0 | 1
Not completed — COPD exacerbation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants (QVA149/Placebo): Participants received 4 weeks of QVA149 and 4 weeks of placebo according to either of the following sequences: QVA149 first and then placebo, or placebo first and then QVA149.
Arm/Group | All Participants (QVA149/Placebo)
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Night-time Blood Oxygenation
Description: The mean night-time blood oxygenation following 4 weeks administration of QVA149 compared to placebo was assessed. Night time oxygenation (SpO2) was measured using polygraphy.
Time Frame: Post 4 weeks administration of QVA149, post 4 weeks administration of placebo
Population: Only randomized participants with data from both treatments were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Oxygenation
Groups:
- QVA149 (Indacaterol/Glycopyrronium); Placebo: Participants received 4 weeks of QVA149 85/43 μg delivered dose once daily in the morning between 08:00 and 11:00 AM at approximately the same time every day.
Arm/Group | QVA149 (Indacaterol/Glycopyrronium) | Placebo
Number analyzed (Participants) | 35 | 34
Percent Oxygenation | 89.59 (0.30) | 90.04 (0.28)
Statistical Analysis 1: Comparison: QVA149 (Indacaterol/Glycopyrronium) vs Placebo; Test type: Superiority or Other; p = 0.2419, Mixed Models Analysis; Mean Difference (Net) = -0.44, 95% CI 2-sided [-1.21 to 0.32]

2. Secondary Outcome: Percent of Time Spent During the Night Below 90 % in Blood Oxygen Saturation
Description: The time during the night spent below 90 % in blood oxygen saturation following 4 weeks administration of QVA149 compared to placebo was assessed. Night time oxygenation (SpO2) was measured using polygraphy.
Time Frame: Post 4 weeks administration of QVA149, post 4 weeks administration of placebo
Population: Only randomized participants with data from both treatments were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | QVA149 (Indacaterol/Glycopyrronium) | Placebo
Number analyzed (Participants) | 35 | 34
Percent | 44.37 (5.09) | 36.58 (4.84)
Statistical Analysis 1: Comparison: QVA149 (Indacaterol/Glycopyrronium) vs Placebo; Test type: Superiority or Other; p = 0.2016, Mixed Models Analysis; Mean Difference (Net) = 7.79, 95% CI 2-sided [-4.51 to 20.08]

ADVERSE EVENTS:
Arm/Group | QVA149 (Indacaterol/Glycopyrronium) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/34
Other Adverse Events (participants affected / at risk) | 14/35 | 12/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (Indacaterol/Glycopyrronium) (N=35) | Placebo (N=34)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (Indacaterol/Glycopyrronium) (N=35) | Placebo (N=34)
Blindness transient (Eye disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2
Blood glucose increased (Investigations) | 0 | 2
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.